CLINICAL TRIAL: NCT05105035
Title: A Randomized, Double-Blind, Placebo-Controlled, Exploratory Study to Assess the Efficacy, Safety and Tolerability of Oral ARV-1801 Given in Combination With Intravenous Ceftazidime or Meropenem for Intensive Phase Therapy of Melioidosis in Hospitalized Patients
Brief Title: Oral ARV-1801 Given in Combination With Intravenous Ceftazidime or Meropenem for Treatment of Melioidosis in Hospitalized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrevus Inc. (Industry)
Collaborators: Arnasi Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARV-1801-001
Record Dates: First submitted 2021-09-23; First posted 2021-11-03 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Melioidosis
Keywords: meropenem; ceftazidime; B. pseudomallei
MeSH Terms: conditions — Melioidosis | interventions — Ceftazidime; Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Active study drug and placebo will appear the same to study staff and patients. Bottles will be blinded to study staff and patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Patients are administered either IV ceftazidime or IV meropenem per standard of care and placebo. Placebo will be administered every 12 hours for Days 1-14.
  Interventions: Drug: Ceftazidime or meropenem; Drug: Placebo
- ARV-1801 (ACG-701) (Experimental): Patients are administered either IV ceftazidime or IV meropenem per standard of care and active ARV-1801. Day 1 dosing will be two doses of 1500mg of ARV-1801 administered 12 hours apart. Days 2-14 dosing will be 600mg of ARV-1801 administered every 12 hours.
  Interventions: Drug: Ceftazidime or meropenem; Drug: ARV-1801

INTERVENTIONS:
Drug: Ceftazidime or meropenem — Patients will be prescribed ceftazidime or meropenem intravenously as per standard of care for at least 14 days while in the hospital
Drug: ARV-1801 — Patients will be prescribed ARV-1801 at 1500mg 12 hours apart on Day 1 and 600mg every 12 hours for Days 2-14.
  Arms: ARV-1801 (ACG-701)
Drug: Placebo — Patients will be prescribed placebo every 12 hours for Days 1-14.
  Arms: Placebo

SUMMARY:
The study investigates the effect of 14 days of twice daily doses of ARV-1801 or placebo in combination with meropenem or ceftazidime in patients hospitalized with melioidosis.

DETAILED DESCRIPTION:
ARV-1801 is an oral dosage form and loading dose regimen of sodium fusidate. Sodium fusidate is a member of the fusidane class of antibiotics. Recent evidence demonstrates meaningful activity against multiple biothreat agents, including the intracellular pathogen B. pseudomallei, which causes melioidosis. Once melioidosis is suspected clinically, treatment typically involves intravenous antibiotics such as ceftazidime or meropenem during an initial "intensive" phase (typically 2 weeks) and oral antibiotics such as co trimoxazole during a more chronic "eradication" phase (typically 12 weeks). Nevertheless, mortality can still exceed 40% in some regions, with most deaths occurring early during the eradication phase of therapy.

The purpose of this study is to evaluate the effects of ARV-1801 administered for 14 days in conjunction with the current standard of care (meropenem or ceftazidime) against placebo in conjunction with the current standard of care. Day 1 dosing will include two doses of 1500mg of ARV-1801 or placebo administered 12 hours apart. Days 2-14 will include 600 mg doses of ARV-1801 or placebo administered every 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must provide written informed consent obtained prior to any study-specific procedure being performed.
2. Patient must be at least 18 years of age or older at time of consent.
3. Patient must be hospitalized with suspected community-acquired melioidosis, meeting at least one of the criteria below:

   * History of frequent contact with soil or surface water in an endemic area
   * Presence of a known underlying risk factor such as diabetes, renal insufficiency, renal stones or thalassemia
   * Special organ involvement such as splenic or hepatic abscess
   * An illness compatible with melioidosis, including the presence of sepsis, acute pneumonia, acute pyelonephritis, septic arthritis, parotid disease or skin or soft tissue infection
4. Patient must require intravenous antibiotics i.e., either ceftazidime or meropenem for treatment of suspected melioidosis.
5. Patient must agree to stay in hospital for duration of ARV-1801 therapy, i.e., 14 days.
6. Females of childbearing potential must use an acceptable method of birth control (surgically sterile, intrauterine device, vasectomized partner, oral contraceptive plus barrier contraceptive, hormone delivery system plus barrier contraceptive or condom in combination with contraceptive cream, jelly or foam) for the duration of the study drug administration phase and for 30 days thereafter.

Exclusion Criteria:

1. Patient is unable to tolerate oral therapy, either directly or via a nasogastric tube.
2. Patient has a known infection with an identified organism other than B. pseudomallei.
3. Patient is pregnant or lactating.
4. Patient has a known hypersensitivity to sodium fusidate, ceftazidime or meropenem.
5. Patient has been treated with IV antibiotics active against B. pseudomallei (including ceftazidime and meropenem) for longer than 48 hours prior to randomization.
6. Patient requires concomitant treatment with the following:

   * OATP1B1 and OATP1B3 substrates, in particular statins (e.g., HMG-CoA reductase inhibitors)
   * Medications metabolized by CYP2C8, such as glitazones (e.g., repaglinide)
   * CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, phenobarbital, and nafcillin)
7. Patient has had prior treatment with a CYP3A4 inducer, such as dexamethasone, phenytoin, carbamazepine, rifampin, phenobarbital, or nafcillin, within 7 days prior to enrollment.
8. Patient requires treatment with digoxin or warfarin unless a monitoring plan is in place to assess digoxin levels and/or prothrombin time as is relevant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
All-cause in-hospital mortality through Day 14 in the modified intent-to-treat population (mITT) | Measured at Day 14

SECONDARY OUTCOMES:
All-cause in-hospital mortality in mITT population | Measured at study completion, on average 28 days (assessed up to 60 days)
All-cause in-hospital mortality through Day 14 in the ITT population | Measured at study completion, on average 28 days (assessed up to 60 days)
All-cause in-hospital mortality in the ITT population | Measured at study completion, on average 28 days (assessed up to 60 days)
Clearance of positive baseline B. pseudomallei blood cultures at Day 1, 3 and 7 | Measured at Days 1, 3 and 7
Number of days in the ICU in the mITT population | Measured at study completion, on average 28 days (assessed up to 60 days)
Number of days on ventilator in the mITT population | Measured at study completion, on average 28 days (assessed up to 60 days)
Length of hospital stay in the mITT population | Measured at study completion, on average 28 days (assessed up to 60 days)
Melioidosis seriousness score in mITT population | Measured at Day 28
Number of patients experiencing adverse events | Measured at study completion, on average 28 days (assessed up to 60 days)

CONTACTS AND LOCATIONS:
Locations (5):
- Thailand (5):
  - Maharat Nakhonratchasima Hospital, Nai Muang
  - Srinagarind Hospital, Khon Kaen University, Nai Muang
  - Sunpasitthiprasong Hospital, Nai Muang
  - Surin Hospital, Nai Muang
  - Udon Thani Hospital, Udon Thani

IPD SHARING:
Plan to Share IPD: No